CLINICAL TRIAL: NCT04306536
Title: Muscle-targeted Nutritional Support in Post-surgical Rehabilitation for Femur Fracture
Brief Title: Nutritional Support in Femur Fracture Rehabilitation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID Pandemic and change in surgical activities in the institution
Sponsor: Barichella Michela (Other)
Responsible Party: Sponsor-Investigator, Barichella Michela, Study coordinator, ASST Gaetano Pini-CTO
Organization: ASST Gaetano Pini-CTO (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: parere 72_2020bis
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Femur Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fortifit® (Experimental): Best local diet + two servings (40 grams each) of powder (Fortifit®; Nutricia) which has to be dissolved in 125 ml of water. Per serving, 20 g whey protein, 3 g total leucine, 9 g carbohydrates, 3 g fat, 800 IU vitamin D, and a mixture of vitamins, minerals, and fibers.
  Interventions: Dietary Supplement: Fortifit®
- Control group (No Intervention): Best local diet

INTERVENTIONS:
Dietary Supplement: Fortifit® — Best local diet + two servings (40 grams each) of powder (Fortifit®; Nutricia) which has to be dissolved in 125 ml of water. Per serving, 20 g whey protein, 3 g total leucine, 9 g carbohydrates, 3 g fat, 800 IU vitamin D, and a mixture of vitamins, minerals, and fibers.
  Arms: Fortifit®

SUMMARY:
This randomized, observer-blinded trial tested the hypothesis that nutritional supplementation with muscle-target nutritional supplementation would increase the efficacy of a physical rehabilitation program in old adults with femur fracture treated with surgery.

DETAILED DESCRIPTION:
Muscle-target nutritional supplementation has been domonstrated to enhance the recovery of muscle mass and increase the efficacy of a rehabilitation program in patients suffering from sarcopenia. Femure fracture is responsible for increased immobilization resulting in loss of muscle mass which may be further emphasized by surgical stress. This randomized, observer-blinded trial tested the hypothesis that nutritional supplementation with muscle-target nutritional supplementation would increase the efficacy of a physical rehabilitation program in old adults with femur fracture treated with surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 60 years or older
* admission for physical rehabilitation after surgery for femur fracture
* informed consent

Exclusion Criteria:

* Any malignant disease during the last five years
* Known kidney failure (previous glomerular filtration rate <30 ml/min);
* Known liver failure (Child B or C)
* Psychiatric disease
* Severe cognitive impairment (Mini Mental State Examination <18)
* Endocrine disorders associated with disorders of calcium metabolism (excluding osteoporosis)
* Indications related to the study product:

  1. More than 10 µg (400 IU) of daily Vitamin D intake from medical sources
  2. More than 500 mg of daily calcium intake from medical sources.
  3. Adherence to a high-energy or high-protein diet (up to three months before starting the study)
  4. Hypersensitivity to any component of the investigational nutritional supplement (including cow milk protein allergy to milk and lactose intolerance)
* Indication to or ongoing artificial nutrition support
* Inclusion in other nutrition intervention trials
* Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* Refusal

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Physical performance - gait speed | 4 weeks
  Gait speed at the 10-meter walking test

SECONDARY OUTCOMES:
Physical performance - Timed Up and Go test | 4 weeks
  Change in timed up and go test
Functional status - Barthel | 4 weeks
  Change in Barthel index score
Functional status - handgrip strength | 4 weeks
  Change in handgrip strength
Body composition - phase angle | 4 weeks
  Change in phase angle
Body composition - muscle mass | 4 weeks
  Change in muscle mass
Body composition - fat-free mass | 4 weeks
  Change in fat-free mass
Body composition - fat-free mass index | 4 weeks
  Change in fat-free mass index
Body weight | 4 weeks
  Change in body weight
Calf circumference | 4 weeks
  Change in calf circumference
Modality of discharge | 4 weeks
  Difference in the proportion of patients discharged at home

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Panella, MD, Principal Investigator — ASST Gaetano Pini-CTO
Locations (1):
- Asst Gaetano Pini, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided